The incidence of chronic non-communicable diseases such as diabetes is increasing with the development of economy and the change of living environment and lifestyle, and it has become one of the major health-threatening diseases. Improper diet is an important cause of metabolic diseases. Reasonable diet can prevent and alleviate such chronic metabolic diseases. Islet dysfunction plays a vital role in the pathophysiological process of diabetes. Therefore, we carried out this survey in order to further understand the relationship between dietary load and islet function, and better promote the prevention, diagnosis and treatment of diabetes.

Subjects are cordially invited to participate in this study with age between 20 to 65 years old, body mass index (BMI, weight [kg] / height [m]<sup>2</sup>) > 18kg/m<sup>2</sup>, and without a history of receiving systemic glucocorticoid therapy for 7 consecutive days in the past 6 months, serious heart, liver, kidney, pancreas and other organ diseases as well as acute or chronic infections.

We will learn about your basic situation, lifestyle and history of chronic diseases through a questionnaire, and will provide you with free oral food (glucose, protein, butter, olive oil or mixed meal tolerance test). Blood sugar, insulin, C-peptide and physical examination will be detected. Blood samples were collected for 5 times with a total volume of 50ml. The process of blood collection may cause pain, stasis, and a very small number of people may have the risk of dizziness of blood or needles, which will generally relieve after rest and do not have health hazards.

We will feedback the test results to you, analyze your metabolic condition and islet function, and provide evaluation for your health status professionally. We will bear the full cost of this inspection. Your personal information and inspection results will be kept confidential and not be disclosed.

PI: Tao Yang

Department: Department of Endocrinology & Metabolism, the First Affiliated Hospital of Nanjing Medical University

## The informed consent signature on a voluntary basis

I have read and learned the information about this health examination. The investigator has fully explained the benefits and losses of the examination, and has given me the opportunity to raise questions. I have gained a satisfactory answer. I agree to participate in this study based on my personal willingness.

| Signature of examinee (or his/her authorized person): |
|-------------------------------------------------------|
| Date: |
| Signature of investigator: |
| Date: |